CLINICAL TRIAL: NCT04961463
Title: Evaluation of the Psychoeducation Program Given to Behcet's Patients in the Context of the Roy Adaptation Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulucanlar Eye Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nermin Erdogan, Principal Investigator, Ulucanlar Eye Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ulucanlar ETRH
Record Dates: First submitted 2021-06-11; First posted 2021-07-14 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Psychoeducation; Nursing Caries; Behcet Syndrome
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Intervention Model Description: The study is a control group quasi-experimental study with a pre-test, post-test and follow-up design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İnterventions group (Experimental): İnterventions group:The 7-session psychoeducation program prepared on the basis of the Roy Adaptation Model was applied to the intervention group once a week for 90-120 minutes
  Interventions: Behavioral: psychoeducation
- Control group (No Intervention): Except for the routine hospital controls, no intervention was made to the control group

INTERVENTIONS:
Behavioral: psychoeducation
  Arms: İnterventions group

SUMMARY:
The physical, social and psychological effects of Behcet's disease necessitate the patient's adaptation in many areas. This study was conducted to examine the effect of psychoeducation given to Behcet's patients in the context of the Roy Adaptation Model on illness adjustment, dyadic adjustment, self-esteem, and psychiatric symptoms. The study is a control group quasi-experimental study with a pre-test, post-test and follow-up design. The study was conducted with 70 Behcet's patients including 35 interventions and 35 controls. The data of the study were collected using the "Patient Information Form", " Adaptation to Chronic Illness Scale", "Dyadic Adjustment Scale", "Rosenberg Self-Esteem Scale" and "Brief Symptom Inventory" in pre-test, post-test and follow-up measurements. A 7-session psychoeducation program was applied to the intervention group.

DETAILED DESCRIPTION:
The research was carried out by using quantitative research methods, quasi-experimental (pre-test, post-test, follow-up, control group) research method.The study was conducted with patients followed-up in eye, dermatology and rheumatology clinics of 6 state-owned hospitals in Ankara, Turkey. The sample size of the study was calculated with the PASS (Power Analysis and Sample Size) statistical package program. It was calculated that our study could be performed with 5% error and 90% power with 35 interventions and 35 control groups, with 70 patients in total. Thus, the research was completed with 70 patients, 35 interventions and 35 control groups.The 7-session psychoeducation program prepared on the basis of the Roy Adaptation Model was applied to the intervention group once a week for 90-120 minutes. Psychoeducation was conducted in 3 groups of 10-12 people, and make-up sessions were held for those who did not attend two consecutive psychoeducation sessions or did not attend two sessions in total. The contents of the psychoeducation sessions were created by the researcher, based on the Roy Adaptation Model, by examining the relevant literature. After the ethics committee report with the permission number GO16 / 229-21 was obtained from the Non-Interventional Clinical Research Ethics Committee of Hacettepe University, the application permission was obtained from the hospitals where the study will be conducted in order to be able to apply the study. Before starting the intervention, the patients were informed about the purpose and scope of the study, and written informed consent was obtained from the patients who agreed to participate in the study. For the control group, after the necessary information was given to the patients, their written informed consent was obtained.

ELIGIBILITY:
Inclusion Criteria:

* Married or had a partner life,
* Were 18 years old

Exclusion Criteria:

* Hearing and speech impairment
* A psychiatric diagnosis
* Neurological involvement

Ages: 23 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of change in disease compliance | 1 week before psychoeducation (pre-test), After the psychoeducation (posttest) and 1 month after posttest
  Adaptation to chronic ilness scale was used to assess disease compliance. The minimum score that can be obtained from the scale is 25 and the maximum score is 125. As the total scale score increases, disease compliance also increases.
Evaluation of change in psychiatric symptoms | 1 week before psychoeducation (pre-test),1 week after the last session of psychoeducation (posttest) and 1 month after posttest
  Brief symptom inventory was used to assess Psychiatric symptoms The minimum score that can be obtained from the scale is 0 and the maximum score is 212. As the total scale score increases, the level of psychiatric symptoms also increases.
Evaluation of change in dyadic adjustment | 1 week before psychoeducation (pre-test),1 week after the last session of psychoeducation (posttest) and 1 month after posttest
  Dyadic adjustment scale was used to assess dyadic adjustment The minimum score that can be obtained from the scale is 0 and the maximum score is 151. Higher total adjustment score indicates better marital adjustment.
Evaluation of change in Self-esteem | 1 week before psychoeducation (pre-test),1 week after the last session of psychoeducation (posttest) and 1 month after posttest
  Rosenberg self-esteem scale was used to assess self-esteem. The minimum score that can be obtained from the scale is 0 and the maximum score is 6. As the total scale score decreases, self-esteem increases

CONTACTS AND LOCATIONS:
Overall Officials: Nermin Erdoğan, Principal Investigator — Ulucanlar Eye Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No